CLINICAL TRIAL: NCT06196827
Title: A Multi-center Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of rAAV2-RPE65 Gene Therapy (LX101) in Subjects With Biallelic RPE65 Mutation-associated Inherited Retinal Dystrophy
Brief Title: Safety and Tolerability of LX101 for Inherited Retinal Dystrophy Associated With RPE65 Mutations
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOSTELLAR-LX101-1 (phase 1)
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Inherited Retinal Dystrophy Associated With RPE65 Mutations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LX101 Dose 1 (Experimental)
  Interventions: Genetic: LX101
- LX101 Dose 2 (Experimental)
  Interventions: Genetic: LX101

INTERVENTIONS:
Genetic: LX101 — Subretinal Administration

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and efficacy of LX101 in subjects with biallelic RPE65 mutation-associated inherited retinal dystrophy.

ELIGIBILITY:
Inclusion Criteria:

Subject and/or their guardian signing a written informed consent.

Diagnosed with biallelic RPE65 mutation-associated inherited retinal dystrophy.

Subjects are 6 years of age or older.

Visual acuity of ≤ 20/63 or visual field less than 20 degrees in the eye to be injected.

Exclusion Criteria:

Prior gene therapy for IRD and other hereditary eye diseases.

Pre-existing eye conditions that would interfere with interpretation of study endpoints.

Active intraocular or periocular infections in the study eye.

Lacking of sufficient surviving retinal cells.

Prior ocular surgery within six months.

Complicating systemic diseases or clinically significant abnormal baseline laboratory values.

Pre-existing systemic diseases that should not discontinue the use of any retinal toxic compounds.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 12 months
  Incidence of ocular and non-ocular AEs and SAEs following LX101 subretinal injection
Incidence of dose-limiting toxicity (DLT) | 1 month
  Incidence of DLT following LX101 subretinal injection at different doses

SECONDARY OUTCOMES:
Efficacy of LX101 in study eye | 12 months
  Changes in BCVA from baseline
Efficacy of LX101 in study eye | 12 months
  Changes in full-field stimulus threshold (FST) from baseline

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Shanghai General Hospital, Shanghai